CLINICAL TRIAL: NCT00928291
Title: The Use of a Procalcitonin (PCT)-Guided Protocol to Shorten the Duration of Antibiotic Therapy in Febrile Neutropenic Patients. An Interventional Study.
Brief Title: Procalcitonin Protocol to Shorten the Antibiotic Therapy in Febrile Neutropenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Vandack Nobre, Associate Professor, PhD
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PCT febrile neutropenia
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2009-12

CONDITIONS: Febrile Neutropenia
Keywords: procalcitonin; neutropenia; febrile neutropenia; antibiotic therapy; neutropenic patients
MeSH Terms: conditions — Febrile Neutropenia; Neutropenia | interventions — Procalcitonin; Anti-Infective Agents

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 - PCT group (Experimental): interventions on antibiotic therapy will be based on circulating PCT levels
  Interventions: Other: procalcitonin; Drug: antibiotic therapy
- Group 2 - Control group (Active Comparator): antibiotic therapy will be guided by appropriate guidelines, and will be left at the discretion of caregivers.
  Interventions: Other: procalcitonin; Drug: antibiotic therapy

INTERVENTIONS:
Other: procalcitonin — plasma PCT measurement
Drug: antibiotic therapy — antibiotic therapy use

SUMMARY:
In this study the investigators aim to test if a procalcitonin (PCT) - guided strategy allows to reduce the antibiotic use in patients with febrile neutropenia hospitalized in a Brazilian tertiary university hospital, causing no harm.

DETAILED DESCRIPTION:
Methods

* Patients and setting: Prospective controlled randomized interventional study of antibiotic therapy in adult with febrile neutropenia.

The study will be conducted in the University Hospital of the Federal University of Minas Gerais, Brazil. This is a 600-bed tertiary hospital, with approximately 1.6 thousands hospitalizations/month. Roughly 120 episodes of febrile neutropenia were recorded in the first semester of 2007, occurring in 100 patients with hematological leucosis or post-BMT. This number rises if one considers other groups of neutropenic patients, such as those with neutropenia due chemotherapy for solid tumors, patients with BM aplasia, myelo dysplasia, among others,

* Interventions:

As long as the core objective of the study is to test if a PCT-guided protocol allows to guide the antibiotic withdrawn in neutropenic patients, only patients with febrile neutropenia under antibiotic therapy will be included in the study. They will be submitted to the following exams:

* Bood samples will be drawn at baseline to blood culture, CRP, blood cells count, ions, liver profile and renal function tests. These exams will be repeated according to the local protocol followed by the Service of Hematology (see appendix).
* A plasma galactomannan test will be performed at baseline in all patients considered for inclusion in the study, and repeated at any moment if there is suspicion of Aspergillus infection during the follow up.
* A chest radiography will also be performed in all participants at baseline, and according to clinical indication afterwards.
* All patients with abnormal chest radiography at baseline will be submitted to a contrasted chest CT (or without contrast if creatinine clearance < 50 ml/min).
* Additional complementary exams will be performed as clinically needed.
* Circulating PCT measurements will be performed at baseline, and then on day 3 (if initial PCT < 0.5) or on day 5 (if initial PCT >0.5).

Eligible patients will be reassessed for on day 3 (if initial PCT < 0.5) or on day 5 (if initial PCT >0.5), and randomized at 1:1 basis to one of the two groups since any exclusion criteria (see below) is present at that time:

Group 1 - PCT group: the interventions on antibiotic therapy will be based on circulating PCT levels.

Group 2 - Control group: antibiotic therapy will be guided by appropriate guidelines, and will be left at the discretion of caregivers.

Patients randomized to the study will undergo daily measurements of plasma PCT levels, and kept under antibiotic therapy until a relative reduction of 90% in baseline PCT levels, or a value lower than 0.5 ng/ml is reached, and then maintained for additional 48h (two measure). Therefore, plasma PCT levels will be measured every 5 days up to the 28th day of follow-up or until death or transference, if either occurs first. Patients included in the interventional group will be observed for at least 48 hours following antibiotic discontinuation before being discharged from the hospital. Extra PCT tests will be performed according to the clinical course.

Apart from the antibiotic therapy, all participants will be managed according to the appropriate guidelines. Patients with febrile neutropenia hospitalized in the University Hospital of the Federal University of Minas Gerais are routinely cared by an experienced hematology specialist together with an infectious diseases consultant. This standard care will be offered to all patients included in the study. The final decision regarding antibiotic therapy will be always let to the discretion of these specialists.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* febrile neutropenia
* to be under antibiotic therapy
* signed informed consent

Exclusion Criteria:

* patients under antibiotic therapy for more than 72 hours before inclusion
* patients post allogenic bone-marrow transplant (BMT)
* patients presenting one or more of the following conditions at the time of randomization:

  * severe mucositis
  * all-trans retinoic acid (ATRA) syndrome
  * disseminated intravascular coagulation
  * hypotension (systolic blood pressure < 90 mmHg or need for vasopressor to maintain blood pressure)
  * respiratory failure (arterial oxygen pressure < 60 mmHg while breathing room air) or need for mechanical ventilation
  * severe renal failure requiring hemodialysis
* patients with suspected (positive galactomannan assay in peripheral blood, nodular lesions with halo in the chest CT) or microbiologically confirmed fungal infection
* bacteremia due to S. aureus
* microbiologically confirmed carbapenem resistant P. aeruginosa or A. baumanii infection
* microbiologically confirmed pneumonia due to P. aeruginosa, A. baumanii or Stenotrophomonas maltophilla
* suspected or confirmed infection caused by atypical microorganisms (virus, parasites, P. jiroveci). Patients with localized HSV infection (e.g., labial) will be accepted for inclusion
* infections requiring prolonged therapies, such as endocarditis and cerebral abscess
* clearly focal bacterial infections

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Antibiotic exposure, measured by: - incidence density of ''antibiotic exposure days'' - incidence rate ratio (IRR) of antibiotic exposure | 28 days
Number of days alive without antibiotics | 28 days
Duration of antibiotic therapy for the first episode of fever | 28 days

SECONDARY OUTCOMES:
Length of hospital stay | 6 m
All cause and infection-related 28-day mortality | 28 days
All cause 90-day mortality | 90 days
Clinical cure rate | 28 days
Nosocomial superinfection (diagnosed more than 48 hours after discontinuation of the antibiotic(s) given to the first episode of infection) | 28 days
Infection relapse (diagnosed less than 48 h after antibiotic discontinuation) | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Vandack Nobre, PhD, Study Chair — Medicine Faculty of Federal University of Minas Gerais; Stella SS Lima, MD, Study Chair — Medicine Faculty of Federal University of Minas Gerais; Henrique NS Bittencourt, PhD, Study Chair — Medicine Faculty of Federal University of Minas Gerais; José C Serufo, PhD, Principal Investigator — Medicine Faculty of Federal University of Minas Gerais
Locations (1):
- Hospital das Clínicas da Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil